CLINICAL TRIAL: NCT06101069
Title: Development of Magnetic Resonance Fingerprinting for Characterization of Brain Tumors After Radiotherapy
Brief Title: Development of MRF for Characterization of Brain Tumors After Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE3323
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor; Brain Necrosis; Brain Metastases; Glioma
Keywords: Magnetic Resonance Fingerprinting; Radiation necrosis
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Contrast Media

STUDY DESIGN:
Intervention Model Description: This is a prospective, observational, multi-cohort, unblinded, single-center study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Volunteer Participants (Experimental): Healthy volunteers will be recruited to evaluate the capability of MRF in conjunction with intravoxel incoherent motion (IVIM) MRI and serve as healthy control data to compare with the participant data.
  Interventions: Procedure: MRF in conjunction with IVIM MRI without contrast
- Participants with Radiation Necrosis (Experimental): The MRI scans (MRF and IVIM) will be performed on participants with newly developed necrosis prior to any further therapy implementation, surgical biopsy, or resection. For the participants undergoing surgical biopsy or resection after the MRI scans, the findings from the analysis of pathological biopsied specimen will serve as pathological confirmation for the MRI imaging findings
  Interventions: Procedure: MRF in conjunction with IVIM MRI without contrast
- Participants with Tumor Recurrence (Experimental): The MRI scans (MRF and IVIM) will be performed on participants with newly developed recurrent prior to any further therapy implementation, surgical biopsy, or resection. For the participants undergoing surgical biopsy or resection after the MRI scans, the findings from the analysis of pathological biopsied specimen will serve as pathological confirmation for the MRI imaging findings
  Interventions: Procedure: MRF in conjunction with IVIM MRI without contrast
- Participants with Brain Metastases (Experimental): The MRI scans (MRF and IVIM) will be performed on participants with newly developed, untreated brain metastases prior to any therapy implementation, surgical biopsy, or resection. For the participants undergoing surgical biopsy or resection after the MRI scans, the findings from the analysis of pathological biopsied specimen will serve as pathological confirmation for the MRI imaging findings
  Interventions: Procedure: MRF in conjunction with IVIM MRI without contrast
- Participants with Primary Gliomas (Experimental): The MRI scans (MRF and IVIM) will be performed on participants with newly developed, untreated primary gliomas prior to any therapy implementation, surgical biopsy, or resection. For the participants undergoing surgical biopsy or resection after the MRI scans, the findings from the analysis of pathological biopsied specimen will serve as pathological confirmation for the MRI imaging findings
  Interventions: Procedure: MRF in conjunction with IVIM MRI without contrast

INTERVENTIONS:
Procedure: MRF in conjunction with IVIM MRI without contrast — MRF in conjunction with IVIM MRI scan, without contrast.

SUMMARY:
The purpose of this study is to discover the potential convenience and ease of using a Magnetic Resonance Imaging (MRI) technique, named Magnetic Resonance Fingerprinting (or MRF), to achieve high-quality images within a short scan time of 5 min for viewing the entire brain. This is an advanced quantitative assessment of brain tissues. This method is being applied with IVIM MRI to be able to tell the difference between a brain with radiation necrosis and a brain with tumor recurrence. Participants will consist of individuals who have received radiation therapy in the past and were diagnosed with radiation necrosis, individuals with recurrent tumors, individuals with previously untreated tumors, and healthy individuals who have no brain diseases and have not had radiation treatment to the brain. Participants will undergo an MRI scan at a one-time research study visit; no extra tests or procedures will be required for this research study.

The primary objectives of this study are:

* To demonstrate the clinical feasibility of combining MRF with state-of-the-art parallel imaging techniques to achieve high-resolution quantitative imaging within a reasonable scan time of 5 min for whole brain coverage.
* To apply the developed quantitative approach in combination with IVIM MRI for differentiation of tumor recurrence and radiation necrosis.
* To investigate the effect of radiation dose on the development of radiation necrosis and tumor recurrence.

DETAILED DESCRIPTION:
Although Stereotactic radiosurgery (SRS) is utilized as an effective treatment method, after several months to over 1 year following SRS, 33% of treated brain metastases increase in size on imaging, which is suspicious for tumor progression. However, based on findings in follow-up biopsies, the majority of newly detected metastases on imaging are radiation treatment effects instead of active tumor. So far, the only gold standard to differentiate active tumor and radiation necrosis is surgical resection for pathologic confirmation, which is invasive, not favored for poor surgical candidates, and should be avoided in cases of necrosis. The existing clinical imaging techniques have poor sensitivity or specificity in differentiating these two types of tissues. Recently, a novel MRI data acquisition approach, namely MR Fingerprinting (MRF), has been introduced for the simultaneous measurement of multiple important parameters in a single MRI scan. In addition, quantitative diffusion MRI, such as the intravoxel incoherent motion (IVIM) technique, can provide a noninvasive and powerful tool to quantify microstructural information by measuring water diffusion and microcirculation perfusion in vivo. This study aims to demonstrate the clinical feasibility of combining MRF with state-of-the-art parallel imaging techniques to achieve high-resolution quantitative imaging within a reasonable scan time of 5 min for whole brain coverage. It also aims to apply the developed quantitative approach in combination with IVIM MRI for the differentiation of tumor recurrence and radiation necrosis. The multi-parametric quantitative measures developed in this study could establish a new fundamental biomarker for the diagnosis and monitoring of brain tumors.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* No history of cerebrovascular disease.
* No cognitive impairments.
* Able to provide informed consent.

Inclusion Criteria for Participants with Brain Tumors:

* Biopsy-proven cases of developed recurrent tumor or radiation necrosis, OR
* a. PET identified with developed recurrent tumor or radiation necrosis. OR
* b. Highly suspicious case with developed recurrent tumor or radiation necrosis confirmed by tumor board, attending physician or surgeon.
* ECOG performance status 0-2.
* Life expectancy > 6 months.
* Participant with other sites of extracranial metastatic disease or any prior or current systemic therapies will be considered and evaluated by the investigators of the study on a subject basis.

Inclusion Criteria for Participants with Brain Metastases or Primary Gliomas:

* Radiology identified with developed primary gliomas tumor or brain metastases, OR
* a. PET identified with developed gliomas tumor or brain metastases, OR
* b. Highly suspicious case with developed gliomas tumor or brain metastases confirmed by tumor board
* Participants must not have received prior radiation or surgical treatment for brain metastases or primary glioma.
* Age: 21 years and over
* ECOG performance status 0-2
* Life expectancy > 6 months.
* Participant with other sites of extracranial metastatic disease or any prior or current systemic therapies will be considered and evaluated by the investigators of the study on a subject basis.

Exclusion Criteria:

* Pregnant women OR lactating women
* Participants with ferromagnetic or otherwise non-MRI compatible aneurysm clips.
* Participants who cannot go into the MRI scanner due to metal implants and other medical conditions.
* The presence of an implanted medical device that is not MRI-compatible, including, but not limited to: pacemaker, defibrillator.
* Participants with contraindications for MRI due to embedded foreign metallic objects such as bullets, shrapnel, metalwork fragments, or other metallic material.
* Known history of severe claustrophobia.
* Participants unable to lay still in the scanner for 30 minutes at a time.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of T1 relaxation times | Within the total 30-45 minute scan time
  The primary objective is to use MRF and IVIM MRI to demonstrate clinical feasibility and differentiation of tumor recurrence and radiation necrosis. This will be measured by the 3D-MRF T1 relaxation times. The difference in mean T1 between each cohort of participants will be measured.
Comparison of T2 relaxation times | Within the total 30-45 minute scan time
  The primary objective is to use MRF and IVIM MRI to demonstrate clinical feasibility and differentiation of tumor recurrence and radiation necrosis. This will be measured by the 3D-MRF T2 relaxation times. The difference in mean T2 between each cohort of participants will be measured.
Comparison of proton density maps | Within the total 30-45 minute scan time
  The primary objective is to use MRF and IVIM MRI to demonstrate clinical feasibility and differentiation of tumor recurrence and radiation necrosis. This will be measured by comparing the MRF proton density maps of each cohort of participants. This will be compared using a t-test.
Comparison of water diffusion in brain tissues | Within the total 30-45 minute scan time
  The primary objective is to use MRF and IVIM MRI to demonstrate clinical feasibility and differentiation of tumor recurrence and radiation necrosis. This will be measured by comparing the diffusion parameters measured by the IVIM method between the three cohorts of participants. This will be compared using a t-test.
Comparison of blood perfusion in brain tissues | Within the total 30-45 minute scan time
  The primary objective is to use MRF and IVIM MRI to demonstrate clinical feasibility and differentiation of tumor recurrence and radiation necrosis. This will be measured by comparing the perfusion parameters measured by the IVIM method between the three cohorts of participants. This will be compared using a t-test.
Comparison of MRF imaging tool in different participant populations | Within the total 30-45 minute scan time
  The objective is to compare the effects of radiation dose on development of radiation and necrosis and tumor recurrence by comparing participants in all cohorts (healthy participants with no brain disease, participants with brain tumors (treated), participants with brain metastases or primary gliomas (previously untreated)). The predictive ability will be assessed by comparing univariable ROC analysis, quantified using area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Lan Lu, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center; Samuel Chao, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No